CLINICAL TRIAL: NCT05730140
Title: Association Between Whole Exon Sequencing and Arterial Stiffness in Patients With Intraoperative Hypotension)
Brief Title: The Association Between the Intraoperative Blood Pressure Changes and Whole Exome Genome
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202209125RINC
Record Dates: First submitted 2023-02-07; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: the Association Between the Arterial Stiffness, Intraoperative Blood Pressure Changes and Genetic Effect

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood sample for whole exome genome
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients undergoing general anesthesia: patients undergoing general anesthesia
  Interventions: Other: this study did not involve interventions; it only observational study

INTERVENTIONS:
Other: this study did not involve interventions; it only observational study — this study did not involve interventions. This study is an observational study for elucidating the intraoperative blood pressure changes, artierial stiffness, and whole exome genome

SUMMARY:
The intraoperative blood pressure changes have been important for postoperative morbidity and mortality. However, some patients did not occur intraoperative hypotension but some patients would have severe intraoperative hypotension. It may be associated with genome related. In this hypothesis, we aim to elucidate the association between the whole exome genome and intraoperaive blood pressure changes.

DETAILED DESCRIPTION:
We aim to elucidate the association between the whole exome genome and intraoperative blood pressure changes.

We will enroll patients older than 20 years old and undergo elective general anesthesia.

Before anesthesia, we will obtain blood sample for whole exome genome test and give arterial line for intraoperative monitor.

After completing surgery, we will follow the patients' all postoperative major organ function.

We hope this study to be able to give us the more information about the specific genetic effect on the arterial stiffness and intraoperative blood pressure changes.

ELIGIBILITY:
Inclusion Criteria:

* elective general surgery

Exclusion Criteria:

* coagulopathy

Ages: 20 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients recieving general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-02-10 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The association between the arterial stiffness and whole exome genome | 15 minutes
  using pearson correlation to describe the association

IPD SHARING:
Plan to Share IPD: No
due to ethical concern